CLINICAL TRIAL: NCT03014024
Title: A Double-blind Placebo-controlled Study of Low-level Laser Therapy After Removal of Cast in Distal Radius Fractures
Brief Title: Low-level Laser Therapy in Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Humaira Sæbø, MS, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016/1633
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Colles' Fracture
Keywords: Distal Radius Fracture; Low Level Laser Therapy
MeSH Terms: conditions — Colles' Fracture; Wrist Fractures | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Level Laser therapy (Experimental): After inclusion in the study, patients will be treated with LLLT. The laser is a super pulsed infrared laser with a wavelength of 904 nm, belonging to laser class 3B. Patient will be treated from dorsal side of the wrist on the fracture area, and distal ulna area from the palmar side. Total 20 second on each side (3 points), with 3,6 J/cm2. the light from the laser is not visible to the eye, and will not give any perceptible stimulus. The x-ray will be used to find the fracture line.
  Interventions: Other: Low-Level Laser Therapy
- Placebo Low-Level Laser therapy (Placebo Comparator): After inclusion in the study, patients will be treated with placebo LLLT. This placebo laser is identical in appearance to the other super pulsed infrared laser with a wavelength of 904 nm, belonging to laser class 3B. Patient will be treated on the same areas, and have the same procedure and time. Since the light from the laser is invisible neither the participant nor the therapist will know whether the laser is a placebo.
  Interventions: Other: Placebo Low Level Laser therapy

INTERVENTIONS:
Other: Low-Level Laser Therapy — The laser is an infrared (invisible) 60 mW 904 nm, made by Irradia Midlaser
  Arms: Low-Level Laser therapy
Other: Placebo Low Level Laser therapy — This i laser is not giving any irradiation, but is identical to the infrared (invisible) 60 mW 904 nm Irradia Midlaser, made by Irradia.
  Arms: Placebo Low-Level Laser therapy

SUMMARY:
Conservative treatment of distal radius fracture is immobilisation with cast for 4-6 weeks. After removing the cast, it is common to still have pain, swelling and reduced mobility in the wrist. The aim of this study is to evaluate the influence of LLLT on the hand.

DETAILED DESCRIPTION:
Patient with distal radius fractures are after removal of the cast are recruited form Bergen Emergency Department, where the are randomly divided into two groups with concealed allocation. Patient will be treated 3 times a week, for 3 week. After removal of the cast, the patients pain threshold, swelling, AROM, strength and function is measured. The patients will meet for following-up controls until 26 weeks after injury.

Changes in outcome measures during the study:

Due to covid 19 virus restrictions, we had to abandon the objective physical measurements as planned. Primary outcome measures were retrieved allowing no physical contact with the participants (Ipad, telephone or e-mail).

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fracture, with or without ulna fracture (Colles' fracture
* The breach must be closed
* after reduction: 0 degrees dorsal displacement of radius
* Under 5 degrees shortening of the radius
* Under 3 mm step in the joint
* 18+ years

Exclusion Criteria:

* People who do not speak Norwegian or English
* If the patient is pregnant
* Patient with Smith fracture
* Wounds over fracture area
* If the patient hav a peripheral neve injury
* If the patient had (previously) operated the wrist
* Persons with verified osteoporosis at the time of injury, systemic inflammatory disease (rheumatism), mental illness, stroke, Parkinson's disease, multiple sclerosis, cancer or congenital malformations in wrist
* If the laser treatment can not be started within 3 days after removal of the cast

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2020-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Function and pain | 26 weeks
  Function will be assessed using Patient Rating Wrist and Hand Evaluation (PRWHE), and questions about night pain/pain killers

SECONDARY OUTCOMES:
Pain assessed using Pressure Algometer | 26 weeks
  Pressure Algometer
Swelling will be assessed using measurement tape | 26 weeks
  Swelling will be assessed using measurement tape
Active range of motion will be assessed using goniometer | 26 weeks
  Active range of motion will be assessed using goniometer
Strength will be assessed using dynamometer | 26 weeks
  Strength will be assessed using dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Jan Magnus Bjordal, Professor, Study Director — University of Bergen
Locations (1):
- Bergen Accident Emergency Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saebo H, Naterstad IF, Joensen J, Stausholm MB, Bjordal JM. Pain and Disability of Conservatively Treated Distal Radius Fracture: A Triple-Blinded Randomized Placebo-Controlled Trial of Photobiomodulation Therapy. Photobiomodul Photomed Laser Surg. 2022 Jan;40(1):33-41. doi: 10.1089/photob.2021.0125. PMID 35030040